CLINICAL TRIAL: NCT06731192
Title: Human Umbilical Cord Mesenchymal Stem Cells for Alport Syndrome: Α Prospective Randomized, Single-blind, Placebo-controlled, Single-center Clinical Trial
Brief Title: Human Umbilical Cord Mesenchymal Stem Cells for Alport Syndrome
Acronym: HUCMSC
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: [2022]00100-3; MR-44-24-042448 (Other Grant/Funding Number: National Health Commission of the People's Republic of China)
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Alport Syndrome
Keywords: Alport syndrome; Human Umbilical Cord Mesenchymal Stem Cells; Randomized Clinical Trial
MeSH Terms: conditions — Nephritis, Hereditary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MSC Theatment (Experimental): Conventional symptomatic supportive treatment and human umbilical cord mesenchymal stem cells treatment
  Interventions: Biological: hUC-MSC
- Placebo Control (Placebo Comparator): Conventional symptomatic supportive treatment and normal saline as a placebo control
  Interventions: Drug: Placebo control drug

INTERVENTIONS:
Biological: hUC-MSC — This group of patients received a total of 2 peripheral intravenous Human umbilical cord mesenchymal stem cells (hUC-MSC) infusions during the treatment period on the basis of conventional symptomatic and supportive treatment. The interval between the two infusions was 14 days, and the single infusion dose was approximately 2×1000,000 cells/Kg.
  Conventional clinical treatment refers to symptomatic treatment with ACEI and ARB drugs.
  Arms: MSC Theatment
Drug: Placebo control drug — This group of patients received a total of 2 intravenous infusions of normal saline (the same volume, specifications and batches used in the experimental group) as a placebo control during the treatment period on the basis of conventional symptomatic and supportive treatment. The interval between the two infusions was 14 days.
  Conventional clinical treatment refers to symptomatic treatment with ACEI and ARB drugs.
  Arms: Placebo Control

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of human umbilical cord mesenchymal stem cells (hUC-MSC) in the treatment of Alport syndrome (AS) in a randomized, single-blind, placebo-controlled trial, to provide a clinical basis for the development of stem cell products for the treatment of AS, and to further clarify the therapeutic effect of hUC-MSC in the treatment of AS.

ELIGIBILITY:
Inclusion Criteria:

* 3 years old ≤Age ≤ 12 years old;
* Meet the diagnostic criteria of Alport syndrome;
* Positive proteinuria or combined hematuria;
* Chronic kidney disease (CKD) stage: I-III stage children, that is, glomerular filtration rate greater than 60 ml/min.1.73m2;
* No history of infectious diseases within 1 week before treatment;
* Negative infectious disease screening;
* No allergic state and related clinical manifestations;
* Signed informed consent (children or their families).

Exclusion Criteria:

* Age <3 years or >12 years old;
* Alport syndrome patients with only microscopic hematuria and normal glomerular filtration rate;
* Patients with significantly reduced renal function, chronic kidney disease stage IV or V, Alport syndrome;
* Patients with other renal diseases;
* Have a history of severe allergic reactions or be allergic to 2 or more foods or drugs;
* Known allergy to stem cells or stem cell-derived products or ingredients in stem cell preparations;
* Have severe heart, liver, lung and other organ dysfunction or have tumors;
* Those with developmental malformations of the urinary system;
* Those with autoimmune diseases and regular use of immunosuppressants;
* Those with serious infectious diseases that are not under control;
* Those with a history of infectious diseases such as HBV, HCV, HIV, syphilis;
* History of surgery or acute trauma or blood loss exceeding 200ml within 3 months;
* Participated in other clinical studies within 3 months;
* Have received any cell product or derivative product treatment within 12 months;
* Other circumstances that the researcher deems inappropriate for inclusion.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Urine protein remission rate | 2 weeks to 12 months after treatment
  Follow-up was performed at 2 weeks, 4 weeks, 6 weeks, 8 weeks, 3 months, 4 months, 5 months, 6 months, 8 months, 10 months, and 12 months after the last hUC-MSC infusion. Urinalysis, 24-hour urine protein quantification, and urine protein/creatinine ratio were tested to evaluate the remission of urine protein after treatment.

SECONDARY OUTCOMES:
Hematuria remission rate | 2 weeks to 12 months after treatment
  Follow-up was performed at 2 weeks, 4 weeks, 6 weeks, 8 weeks, 3 months, 4 months, 5 months, 6 months, 8 months, 10 months, and 12 months after the last hUC-MSC infusion. The urine abnormal red blood cell count of the children was tested to evaluate the remission of hematuria after treatment.
Renal function improvement rate | 2 weeks to 12 months after treatment
  Follow-up was performed at 2 weeks, 4 weeks, 6 weeks, 8 weeks, 3 months, 4 months, 5 months, 6 months, 8 months, 10 months, and 12 months after the last hUCMSC infusion to measure the serum creatinine, blood urea nitrogen, serum cystatin C, glomerular filtration rate and other indicators of the children to evaluate the improvement of renal function after treatment.

IPD SHARING:
Plan to Share IPD: No